CLINICAL TRIAL: NCT03641157
Title: Value of BMI and Anthropometric Measurements With CL Test in Predicting Difficult Laryngoscopy in Children
Brief Title: Predicting Difficult Airway in Children
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, GAYE AYDIN, Anesthesiology and Reanimation Clinic, principal investigator, Clinical Associated Professor, Tepecik Training and Research Hospital
Other Study IDs: GAYDIN
Record Dates: First submitted 2018-03-31; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Difficult Intubation; Pediatrics
Keywords: Difficult intubation; Pediatrics; predictive tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I Easy Intubation: Pediatric patients ages 0-3 years Easy Intubation (Cormach-Lehane score I-II)
  Interventions: Other: Easy Intubation
- Group II Difficult intubation: Pediatric patients ages 0-3 years Difficult intubation (Cormach-Lehane score III-IV)
  Interventions: Other: Easy Intubation

INTERVENTIONS:
Other: Easy Intubation
  Other Names: Difficult intubation

SUMMARY:
Background: Obtaining airway security holds the utmost importance in anesthesia. Specific predictive tests or findings for difficult airway are not defined for various pediatric age groups. Anthropometric measurements are defined parallel to percentile curves in different age groups.

Aim: The aim of this study is to find out the value of body mass index and anthropometric measurements in prediction of difficult laryngoscopy in children by comparing to direct laryngoscopic evaluation of Cormack-Lehane test.

Methods: Following institutional ethics committee approval and informed consent of parents of 108 patients (ages 0-3years), undergoing elective surgery were included in this study. Weight, height, body mass index and head circumference of the patients were measured and percentiles were recorded, prior to induction.

Following standard anesthesia induction with thiopental all patients received 0,6 mg.kg-1 rocuronium intravenously. After sufficient time for neuromuscular relaxation laryngoscopy performed and Cormack-Lehane scores recorded. All recorded parameters were compared with Cormack-Lehane scores.

ELIGIBILITY:
Inclusion Criteria:

* 0-3 years old (1-36 mounts) pediatric patients
* Patients 0-3 age years old with ASA I, undergoing elective surgery were included in this study

Exclusion Criteria:

* Patients with known syndrome, facial anomaly, ASA score above 2 and laryngeal mask aiway were excluded from the study

Ages: 1 Month to 36 Months | Sex: All
Age Groups: Child
Gender Based: Yes — pediatric patients
Study Population: Demographic data, head circumference, weight, height measurements, body mass index and percentile values were recorded by a pediatric surgeon who was unaware about the studyin the preoperative period.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2014-07-11 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2016-07-11 (Actual)

PRIMARY OUTCOMES:
Difficult laryngoscopy classification using Cormack-LehaneGrade Assessment of difficult laryngoscopy at the time of the airway management procedure. | immediate
  Classified as Grade I-visualization of entire laryngeal aperture, grade II-visualization of only posterior commissure of laryngeal aperture, grade III-visualization of only epiglottis, grade IV-visualization of just the soft palate.

SECONDARY OUTCOMES:
Head circumference measured in cm with a measuring tape. | immediate
  Head circumference were taken at the level above eyebrows and ears and measured in cm with a measuring tape.
Weight measured in kilogram with electronic scale. | immediate
  Weight measured using electronic scale (0-20 kg) while undressed and without diapers .
Height measured in cm with infantometer. | immediate
  Height measured using a portable infantometer (0-100 cm) while the child was in supine position.
BMI was calculated as kg/m2. | immediate
  BMI measured using a weight/height2 formul
Percentage values measured in % with percentile tables. | immediate
  Percentage (%) values using from the percentile tables of Turkish children were determined after the head circumference (cm), height (cm), weight (kg) and BMI (kg/m2) values of all pediatric cases were determined as described above.

CONTACTS AND LOCATIONS:
Overall Officials: PERVIN BOZKURT, Prof, Study Director — Tepecik Education and Research Hospital
Locations (1):
- Tepecik Education and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Value of BMI and Anthropometric Measurements with CL Test in Predicting Difficult Laryngoscopy in Children

REFERENCES:
- [Result] Heinrich S, Birkholz T, Ihmsen H, Irouschek A, Ackermann A, Schmidt J. Incidence and predictors of difficult laryngoscopy in 11,219 pediatric anesthesia procedures. Paediatr Anaesth. 2012 Aug;22(8):729-36. doi: 10.1111/j.1460-9592.2012.03813.x. Epub 2012 Feb 20. PMID 22340664
- [Result] Heinrich S, Birkholz T, Ihmsen H, Irouschek A, Ackermann A, Cesnjevar R, Schmidt J. Incidence and predictors of poor laryngoscopic view in children undergoing pediatric cardiac surgery. J Cardiothorac Vasc Anesth. 2013 Jun;27(3):516-21. doi: 10.1053/j.jvca.2012.08.019. Epub 2012 Oct 17. PMID 23083795
- [Result] Inal MT, Memis D, Sahin SH, Gunday I. [Comparison of different tests to determine difficult intubation in pediatric patients]. Rev Bras Anestesiol. 2014 Nov-Dec;64(6):391-4. doi: 10.1016/j.bjan.2014.02.001. Epub 2014 Aug 28. Portuguese. PMID 25437694
- [Result] Mansano AM, Modolo NS, Silva LM, Ganem EM, Braz LG, Knabe Ade C, Freitas FM. Bedside tests to predict laryngoscopic difficulty in pediatric patients. Int J Pediatr Otorhinolaryngol. 2016 Apr;83:63-8. doi: 10.1016/j.ijporl.2016.01.031. Epub 2016 Feb 3. PMID 26968055
- [Result] Mirghassemi A, Soltani AE, Abtahi M. Evaluation of laryngoscopic views and related influencing factors in a pediatric population. Paediatr Anaesth. 2011 Jun;21(6):663-7. doi: 10.1111/j.1460-9592.2011.03555.x. Epub 2011 Mar 14. PMID 21401798